CLINICAL TRIAL: NCT01531738
Title: Investigation of the Effects of Bariatric Surgery on Taste Reward in Humans
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Carel Le Roux, Principal Investigator, Imperial College London
Other Study IDs: PRT
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Taste; bariatric surgery; food preferences; reward; progressive ratio task
MeSH Terms: conditions — Obesity; Food Preferences

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Normal weight healthy volunteers
- Bariatric Surgery: obese patients due to undergo gastric bypass or gastric banding

SUMMARY:
The investigators hypothesize that some of these changes in the reduced appetite after surgery may be due to alterations in taste. The aim is to compare obese patients before and after bariatric surgery (gastric bypass and banding) to define the reward value of sweet, fatty and vegetable/fruit taste in obese individuals, and how this changes after surgery.

DETAILED DESCRIPTION:
Severe obesity is associated with excessive food eating and appetite. Bariatric surgery (also known as 'obesity surgery' or 'weight loss surgery') is a well known treatment for severely obese individuals. The way in which these operations achieve weight loss is not fully understood. The investigators hypothesize that some of these changes in the reduced appetite after surgery may be due to alterations in taste. The aim is to compare obese patients before and after bariatric surgery (gastric bypass and banding) to define the reward value of sweet, fatty and vegetable/fruit taste in obese individuals, and how this changes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-25 for normal weight volunteers
* BMI of >30 for obese patients

Exclusion Criteria:

* Pregnancy
* breast feeding
* substance abuse
* consumption of more than 3 alcoholic units per day
* severe psychiatric illness
* lack of understanding of test instructions
* diabetes mellitus
* chronic medical conditions making a general anaesthetic unsafe
* allergy to stimulus ingredients
* active smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obesity attending a specialist obesity clinic and normal weight controls who are staff at Imperial College London
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel W le Roux, MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Weight Centre, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miras AD, Jackson RN, Jackson SN, Goldstone AP, Olbers T, Hackenberg T, Spector AC, le Roux CW. Gastric bypass surgery for obesity decreases the reward value of a sweet-fat stimulus as assessed in a progressive ratio task. Am J Clin Nutr. 2012 Sep;96(3):467-73. doi: 10.3945/ajcn.112.036921. Epub 2012 Jul 25. PMID 22836034

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Bariatric Surgery
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Bariatric Surgery | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 39 (5) | 49 (3) | 44 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
BMI ("kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 23 (1) | 48 (2) | 35.5 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Breakpoints as Assessed by Change in the Number of Mouse Clicks in the Last Completed Ratio
Description: Patients were placed in front of a computer screen and a plate of 20 chocolate candies. The following prompt appeared on the screen: "You can earn food by clicking on the mouse button. Click as much or as little as you like. When you no longer want to continue, press the spacebar to stop the session."Upon completion of each ratio a message box appeared on the screen: "You have earned food. Enjoy your reward and after you have swallowed it completely you may click on OK to continue with the programme."After ingesting the reward, the patients pressed the OK button in the message box only if they wished to progress to the next ratio to obtain another chocolate candy. The starting ratio was 10 clicks with a geometric increment of 2 (i.e., 10, 20, 40, 80, and so on). When the effort of pressing the mouse button was greater than the rewarding value of the chocolate candy, patients pressed on the space bar to terminate the session. This indicated that the breakpoint was reached.
Time Frame: 2 weeks pre and 8-12 weeks post operatively for surgical patients or on two occasions 10-14 weeks apart for normal weight control group
Measure: Mean (Standard Deviation); unit: Clicks
Arm/Group | Control | Bariatric Surgery
Number analyzed (Participants) | 11 | 11
Clicks | 0 (40) | 320 (30)

2. Secondary Outcome: Hunger
Description: Visual Analogue Scale ratings of hunger. The scale is 100mm line with two anchors at each end. Scores are recorded by making a handwritten mark that represents a continuum between "not hungry at all" and "Extremely hungry." The score of 0 represents least hunger. The score of 100 represents extreme hunger.
  change in hunger levels quantified by a 100mm visual analogue scale
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control | Bariatric Surgery
Number analyzed (Participants) | 11 | 11
mm | 20 (30) | -60 (30)

3. Secondary Outcome: Body Mass Index
Description: change in BMI will be quantified based on the participants weight in kilograms and height in meters
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control | Bariatric Surgery
Number analyzed (Participants) | 11 | 11
kg/m^2 | -0.2 (1.2) | -6.2 (1.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Bariatric Surgery
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes